CLINICAL TRIAL: NCT01855659
Title: A Single-center Study to Assess Peak Inspiratory Flow (PIF) in Different Stages' COPD Patients by Using the In-check Method.
Acronym: INSPIRE
Status: Completed | Type: Observational
Sponsor: Elpen Pharmaceutical Co. Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2013-HAL-EL-36
Record Dates: First submitted 2013-05-14; First posted 2013-05-16 (Estimated); Last update posted 2013-12-03 (Estimated); Status verified 2013-05

CONDITIONS: Pulmonary Disease
Keywords: Lung diseases,; Obstructive,; Peak Inspiratory Flow; [C08.381.495.389]
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- COPD patients: Patients who are stratified in the subgroups of COPD based on the severity: stages II, III, IV

SUMMARY:
Peak Inspiratory Flow Rate (PIFR) is defined by the fastest flow rate noted during the inspiratory cycle.

Inhaled medication plays an important role in the treatment of chronic obstructive pulmonary disease (COPD), with dry powder inhalers (DPIs) increasingly replacing metered dose inhalers (MDIs). DPIs are interesting as they do not require the need for coordinate actuation of the MDI device with inhalation or the use of a large spacer device 1-3. Several DPIs are available for the administration of inhaled corticosteroids, as well as bronchodilators, with each of them corresponding to a different type of inhaler (e.g. Diskus®, Turbuhaler®, Aeroliser®, etc.). During the inspiratory effort the patient generates a pressure drop with a consequent airflow across the DPI. This inspiratory flow has to be high enough to disaggregate and adequately disperse the drug powder into an aerosol cloud of drug particles and to guarantee an optimal deposition of the medication in the lung. Such peak inspiratory flows (PIFs) are not only dependent on a patient's inhalation effort but also on the internal resistance of the device.

It has been shown that optimal deposition of medication with DPIs is not achieved in some patients with low inspiratory flow rates, such as children or patients with COPD, especially during acute exacerbations. In such conditions the use of a DPI with low internal resistance has been suggested, ensuring an optimal deposition despite the lower flow rate. In addition, many clinicians are nowadays confronted with an important number of COPD patients who are aged >70 yrs

DETAILED DESCRIPTION:
This study will assess the inspiratory flow rates at high levels of resistance in different stages of COPD patients. PIF will be measured by in-check method.

Commonly used for Asthma patients, the In-Check Oral Inspiratory Flow Meter is a portable hand-held inspiratory flow meter that provides an assessment of the speed of inhalation. The In-Check Oral measures inspiratory flow between 30 and 370 L/min, inspiratory flow is thought of by physicians as a sensitive marker for Chronic Obstructive Pulmonary Disease (COPD) screening. The In-Check Oral works when a patient inhales through the mouth, this will cause air to be drawn through the meter and a cursor moves along the scale to indicate the speed of inhalation. The flow rate achieved can be noted by checking the position of the cursor against the calibrated scale. The Standard In-Check Oral inspiratory flow meter can measure inspiratory flow rates in the range 30 to 370 l/min, with an accuracy of +/- 10% or 10 l/min (whichever is the greater). (A Low Range In-Check Oral Inspiratory flow meter is available by special request, measuring between 15 and 120 l/min).

All In-Check Oral meters are calibrated using an ATS pulmonary waveform generator, and the product complies with the Australian and New Zealand standards for back pressure in flow meters. As with any inhalation device checking for loose foreign objects is important. The transparent body of the In-Check Oral meter is designed to allow a visual inspection before use. The meter is manufactured from medical grade components, and is suitable for multiple patient uses when cleaned appropriately between patients. The expected life of the In-Check Oral, in normal use, is two years.

Commonly used for Asthma patients, the In-Check Oral Inspiratory Flow Meter is a portable hand-held inspiratory flow meter that provides an assessment of the speed of inhalation. The In-Check Oral measures inspiratory flow between 30 and 370 L/min, inspiratory flow is thought of by physicians as a sensitive marker for Chronic Obstructive Pulmonary Disease (COPD) screening. The In-Check Oral works when a patient inhales through the mouth, this will cause air to be drawn through the meter and a cursor moves along the scale to indicate the speed of inhalation. The flow rate achieved can be noted by checking the position of the cursor against the calibrated scale. The Standard In-Check Oral inspiratory flow meter can measure inspiratory flow rates in the range 30 to 370 l/min, with an accuracy of +/- 10% or 10 l/min (whichever is the greater). (A Low Range In-Check Oral Inspiratory flow meter is available by special request, measuring between 15 and 120 l/min).

All In-Check Oral meters are calibrated using an ATS pulmonary waveform generator, and the product complies with the Australian and New Zealand standards for back pressure in flow meters. As with any inhalation device checking for loose foreign objects is important. The transparent body of the In-Check Oral meter is designed to allow a visual inspection before use. The meter is manufactured from medical grade components, and is suitable for multiple patient use when cleaned appropriately between patients. The expected life of the In-Check Oral, in normal use, is two years.

Commonly used for Asthma patients, the In-Check Oral Inspiratory Flow Meter is a portable hand-held inspiratory flow meter that provides an assessment of the speed of inhalation. The In-Check Oral measures inspiratory flow between 30 and 370 L/min, inspiratory flow is thought of by physicians as a sensitive marker for Chronic Obstructive Pulmonary Disease (COPD) screening. The In-Check Oral works when a patient inhales through the mouth, this will cause air to be drawn through the meter and a cursor moves along the scale to indicate the speed of inhalation. The flow rate achieved can be noted by checking the position of the cursor against the calibrated scale. The Standard In-Check Oral inspiratory flow meter can measure inspiratory flow rates in the range 30 to 370 l/min, with an accuracy of +/- 10% or 10 l/min (whichever is the greater). (A Low Range In-Check Oral Inspiratory flow meter is available by special request, measuring between 15 and 120 l/min).

* All In-Check Oral meters are calibrated using an ATS pulmonary waveform generator, and the product complies with the Australian and New Zealand standards for back pressure in flow meters. As with any inhalation device checking for loose foreign objects is important. The transparent body of the In-Check Oral meter is designed to allow a visual inspection before use. The meter is manufactured from medical grade components, and is suitable for multiple patient use when cleaned appropriately between patients. The expected life of the In-Check Oral, in normal use, is two Accurately measures oral inspiratory flow rate (peak and sub-maximal) in order to assess suitability for inhaled medication
* Measures nasal inspiratory flow for assessing nasal airway patency
* Assesses response to nasal provocation
* Allows home monitoring of Peak Nasal Inspiratory Flow (PNIF)
* Easy to use, clean and reset, the In-Check helps patients maintain their respiratory health.
* High-quality medical-grade stainless steel and plastic construction
* Sterilizable plastic mouthpiece accepts different mask sizes
* Simple enough for home patient use, rugged enough for routine clinic use.

ELIGIBILITY:
Inclusion Criteria:

* COPD patients (Global Initiative of Chronic Lung Disease (GOLD) definition
* COPD stage II, III, IV
* Patients who are followed in Outpatients' Unit
* Patients >50 years of age
* Patients who accept PIF to be measured using the In-Check Inhaler
* Patients who have signed the Informed Consent
* Patients who will comply with study demands and procedures

Exclusion Criteria:

* COPD stage I patients
* Patients who are hospitalized
* Patients <50 years of age
* Patients who do not accept PIF to be measured using the In-Check Inhaler
* Patients who have not signed the Informed Consent
* Patients who face problems in order to comply with study demands and procedures

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD patients belonging in Stages II, II, IV
Sampling Method: Non-Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2013-06; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
PIF measurements in COPD | 0 (baseline)
  Values of PIF measurement in COPD stages' subgroups

SECONDARY OUTCOMES:
PIF measurement in COPD per age and gender | 0 (baseline)
  Values of PIF measurement in COPD patients per age and gender

CONTACTS AND LOCATIONS:
Overall Officials: Eleftherios Zervas, M.D, Study Chair — Coordinator of Asthma Working Group of Hellenic Thoracic Society
Locations (1):
- 7th Pulmonary Dept, Athens Chest Hospital, Athens, Mesogion Ave. 152, Greece

REFERENCES:
- [Background] Melissinos CG, Mead J. Maximum expiratory flow changes induced by longitudinal tension on trachea in normal subjects. J Appl Physiol Respir Environ Exerc Physiol. 1977 Sep;43(3):537-44. doi: 10.1152/jappl.1977.43.3.537. PMID 914724
- [Background] Malik SK, Jindal SK, Jindal V, Bansal S. Peak expiratory flow rate in healthy adults. Indian J Chest Dis. 1975 Oct;17(4):166-71. No abstract available. PMID 1218939
- [Background] Potter WA, Olafsson S, Hyatt RE. Ventilatory mechanics and expiratory flow limitation during exercise in patients with obstructive lung disease. J Clin Invest. 1971 Apr;50(4):910-9. doi: 10.1172/JCI106563. PMID 5547281
- [Background] Schwela D. Air pollution and health in urban areas. Rev Environ Health. 2000 Jan-Jun;15(1-2):13-42. doi: 10.1515/reveh.2000.15.1-2.13. PMID 10939084
- [Background] Singh V, Khandelwal R, Gupta AB. Effect of air pollution on peak expiratory flow rate variability. J Asthma. 2003 Feb;40(1):81-6. doi: 10.1081/jas-120017210. PMID 12699215
- [Background] Njoku CH, Anah CO. Reference values for peak expiratory flow rate in adults of African descent. Trop Doct. 2004 Jul;34(3):135-40. doi: 10.1177/004947550403400303. PMID 15267038
- [Background] Quanjer PH, Lebowitz MD, Gregg I, Miller MR, Pedersen OF. Peak expiratory flow: conclusions and recommendations of a Working Party of the European Respiratory Society. Eur Respir J Suppl. 1997 Feb;24:2S-8S. No abstract available. PMID 9098701
- [Background] Elebute EA, Femi-Pearse D. Peak flow rate in Nigeria: anthropometric determinants and usefulness in assessment of ventilatory function. Thorax. 1971 Sep;26(5):597-601. doi: 10.1136/thx.26.5.597. PMID 5134061
- [Background] Onadeko BO, Iyun AO, Sofowora EO, Adamu SO. Peak expiratory flow rate in normal Nigerian children. Afr J Med Med Sci. 1984 Mar-Jun;13(1-2):25-32. PMID 6087636